CLINICAL TRIAL: NCT06824259
Title: The Value of Dual-parametric Magnetic Resonance Combined With Regional Saturation Biopsy in Diagnostic Decision-making in Patients With Suspected Prostate cancer--a Single-center Prospective Randomized Controlled Study
Brief Title: The Value of Dual-parametric Magnetic Resonance Combined With Regional Saturation Biopsy in Patients With Suspected Prostate Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: bpMRIRSB
Record Dates: First submitted 2025-02-05; First posted 2025-02-13 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MRI negative without biopsy (Experimental): If a lesion with a PI-RADS score of 3 or higher was identified during the initial examination, a regional saturation biopsy of the prostate was conducted, as clinical suspicion of prostate cancer had been raised. Should the initial prostate biopsy yield negative results, the patient would be placed in the follow-up cohort. Targeted biopsy in conjunction with a 12-needle systematic biopsy would only be performed in cases where there was high suspicion of MRI persistence (a PI-RADS v2.1 score of 4 or 5) or if the lesion showed signs of progression. If no lesions with a PI-RADS v2.1 score of 3 or higher were detected during the initial examination, the patients would be entered into the follow-up cohort. Reginal saturation biopsy would be performed when MRI showed progression. If the initial prostate biopsy was negative, the patient would again be entered into the follow-up cohort.
  Interventions: Procedure: Follow up if MRI is negative
- MRI negative with systemic biopsy (Active Comparator): Focal saturation biopsy of the prostate was performed if a PI-RADS v2.1 score ≥3 lesion was detected during the initial examination. If no PIRADS v2.1 score ≥3 lesions were identified, a 12-needle systematic biopsy was performed. If the initial prostate biopsy was negative for prostate cancer, it was entered into the follow-up cohort. When the following clinical indications for repeat biopsy were met ① initial biopsy pathology showed no evidence of malignancy, but atypical small follicular hyperplasia was found, or high-grade epithelial neoplasia in more than 3 needles, with atypical glands visible in the surrounding area present; ② review of persistent elevation of serum PSA or abnormalities in the imaging follow up; and ③ review of serum PSA 4~10 ng/ml in conjunction with f/t PSA, PSAD, PSAV, and PHI, abnormal rectal digital examination or other imaging findings, then target biopsy combined with 12-needle systemic biopsy was performed.
  Interventions: Procedure: Systematic biopsy if MRI is negative

INTERVENTIONS:
Procedure: Follow up if MRI is negative — Enter the follow-up cohort without systematic biopsy when prostate cancer is clinically suspected and no PIRADS v2.1 score ≥3 lesions are detected on initial examination. MR plus regional saturation biopsy was performed when MRI progressed.
  Arms: MRI negative without biopsy
Procedure: Systematic biopsy if MRI is negative — Systematic biopsy was performed if there was clinical suspicion of prostate cancer and no PIRADS v2.1 score ≥3 lesions were detected on initial examination. If the biopsy was negative enter the follow-up cohort.
  Arms: MRI negative with systemic biopsy

SUMMARY:
The aim of this study was to investigate the value of dual-parameter magnetic resonance imaging(bpMRI) combined with regional saturation biopsy in the diagnosis of prostate cancer by means of a prospective randomized controlled study.

The main questions it aims to answer are:

Can bpMRI guide the timing of prostate puncture and avoid unnecessary prostate biopsy? Effectiveness of focal saturation biopsy versus systemic biopsy + targeted biopsy.

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 years of age or older.
2. Compliance with clinical guidelines for indications for prostate puncture:

   * suspicious prostate nodule detected on rectal palpation;
   * suspicious lesion detected by transrectal ultrasound or magnetic resonance;
   * tPSA > 10 ng/mL;
   * tPSA 4-10 ng/mL with f/t < 0.16 or PSAD > 0.15.
3. Complete sequence of bpMRI of the prostate at our institution;

Exclusion Criteria:

1. tPSA >50ng/mL;
2. Presence of contraindications to prostate puncture and inability to tolerate prostate puncture;
3. reatment with radiotherapy, chemotherapy and surgery before prostate puncture;
4. History of prostate cancer;
5. Prostate multiparametric magnetic resonance images of poor quality or some sequences are missing.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
The clinically significant prostate cancer (csPCa) detection rate | One month after the biopsy procedure.
  csPCa was defined as PCa with a grade group > 2 or GS ≥ 7. The reference standard was the pathological result.

SECONDARY OUTCOMES:
The Gleason score (GS) of the biopsy sample | One month after the biopsy procedure.
  The Gleason score (GS) was reported by senior uropathologists according to the Standards of Reporting for MRI Targeted Biopsy Studies (START) criteria and interpreted according to the recommendations of the International Society of Urological Pathology (ISUP) Grade Group. The minimum and maximum of GS are 3 and 5. The higher GS means the higher pathological grade.
The PCa detection rate | One month after the biopsy procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China